CLINICAL TRIAL: NCT06649162
Title: A Multi-center, Prospective, Cohort Study to Identify the Risk of Non-alcoholic Fatty Liver Disease (NAFLD) in Patients With Type 2 Diabetes in Clinical Practice and to Evaluate the Clinical Usefulness of Dapagliflozin/Pioglitazone Combination Therapy
Brief Title: A Study to Identify the Risk of Non-alcoholic Fatty Liver Disease (NAFLD) in Patients With Type 2 Diabetes in Clinical Practice and to Evaluate the Clinical Usefulness of Dapagliflozin/Pioglitazone Combination Therapy
Status: Recruiting | Type: Observational
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: BR-DPC-OS-401
Record Dates: First submitted 2024-10-17; First posted 2024-10-18 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to identify the risk of non-alcoholic fatty liver disease (NAFLD) in patients with type 2 diabetes in clinical practice and to evaluate the clinical usefulness of Dapagliflozin/Pioglitazone combination therapy

ELIGIBILITY:
Inclusion Criteria:

* Among patients with type 2 diabetes, those who are scheduled to administer a fixed-dose combination of dapagliflozin/pioglitazone at baseline (visit 1)
* Those who voluntarily signed a written personal information collection and usage agreement after listening to an explanation about the objective and method, etc. of this clinical study.

Exclusion Criteria:

* Those who have a history of taking a fixed-dose combination of dapagliflozin/pioglitazone at baseline (visit 1).
* Those who are expected to need insulin prescription during the study period.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with type 2 diabetes scheduled to administer a fixed-dose combination of dapagliflozin/pioglitazone
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects who correspond to high risk score (≥8) by evaluating simple NAFLD score | Baseline (visit 1)

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Andong Hospital, Andong, Gyeongsangbuk-do
  - Konkuk University medical center, Seoul

IPD SHARING:
Plan to Share IPD: No